CLINICAL TRIAL: NCT07286214
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Each of Two Dose Levels of Sarilumab in Adults With Early Polymyalgia Rheumatica
Brief Title: Sarilumab Efficacy and Safety in Adults With Early Polymyalgia Rheumatica
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC18055; 2024-511296-15-00 (EU CTIS Number); U1111-1310-5173 (Registry Identifier: ICTRP)
Record Dates: First submitted 2025-12-10; First posted 2025-12-16 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Polymyalgia Rheumatica
MeSH Terms: conditions — Polymyalgia Rheumatica | interventions — sarilumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants will receive placebo with prednisone taper
  Interventions: Drug: Placebo
- Sarilumab 150 mg (Experimental): Participants will receive 150 mg sarilumab q2w with prednisone taper
  Interventions: Drug: Sarilumab
- Sarilumab 200 mg (Experimental): Participants will receive 200 mg sarilumab q2w with prednisone taper
  Interventions: Drug: Sarilumab

INTERVENTIONS:
Drug: Sarilumab — Pharmaceutical form: Solution for injection - Route of administration: Subcutaneous
  Other Names: Kevzara®
  Arms: Sarilumab 200 mg
Drug: Sarilumab — Pharmaceutical form: Solution for injection - Route of administration: Subcutaneous
  Other Names: Kevzara®
  Arms: Sarilumab 150 mg
Drug: Placebo — Pharmaceutical form: Solution for injection - Route of administration: Subcutaneous
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, parallel-group, Phase 4, 3-group study to assess whether treatment with sarilumab at either 150 mg q2w (once every two weeks) or at 200 mg q2w, each given with a 52-week prednisone taper, is superior to placebo given with a 52-week prednisone taper in participants with early polymyalgia rheumatica (PMR) and to determine the safety and tolerability of the sarilumab regimens.

The study will consist of the following visits:

Visit 1 (D-42 to D-1): Screening, Visit 2 (D1): Baseline, randomization, first study drug administration, Visit 3 to 12 (Week 2 to Week 52): Treatment period, Visit 13 (Week 52): End of Treatment (EOT) visit, Visit 14 (Week 58): End of Study (EOS) visit.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥50 years with polymyalgia rheumatica according to the EULAR/ACR classification criteria
* Meet criteria for newly diagnosed PMR (received ≤6 weeks of corticosteroids prior to randomization) or for early relapsing PMR (initiated corticosteroid treatment within last year, treated with prednisone ≥10 mg/day for ≥ 8 weeks, and experienced flare within prior 12 weeks while receiving ≥5 mg/d prednisone)
* Participants must be willing and able to take prednisone of 15 mg/day at randomization
* Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies

Exclusion Criteria:

* Diagnosis of Giant Cell Arteritis (GCA)
* Concurrent rheumatoid arthritis, inflammatory arthritis, connective tissue diseases, fibromyalgia
* Inadequately treated hypothyroidism
* Exclusion related to tuberculosis (TB), invasive opportunistic infections, recurrent or persistent infections including hepatitis B, C or HIV, recurrent herpes zoster or active herpes zoster
* Patients with uncontrolled diabetes mellitus (HbA1c ≥9%)
* Immunosuppressive therapies including systemic corticosteroids
* Malignancy
* Organ transplant recipient

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2026-04-15 (Estimated); Primary Completion 2029-06-04 (Estimated); Study Completion 2029-07-16 (Estimated)

PRIMARY OUTCOMES:
Sustained remission at Week 52 (yes/no) in participants with early relapsing polymyalgia rheumatica (PMR) who received sarilumab 200 mg q2w with 52-week prednisone taper | at Week 52
  No signs or symptoms of PMR at Week 24 and sustained through week 52 (without use of rescue therapy).

SECONDARY OUTCOMES:
Sustained remission at Week 52 (yes/no) in all participants (newly diagnosed PMR and early relapsing PMR) who received sarilumab 200 mg q2w with prednisone taper | at Week 52
  No signs or symptoms of PMR at Week 24 and sustained through week 52 (without use of rescue therapy).
Sustained remission at Week 52 (yes/no) in participants with early relapsing PMR, as well as in all participants (newly diagnosed PMR and early relapsing PMR) who received sarilumab 150 mg q2w with prednisone taper | at Week 52
  No signs or symptoms of PMR at Week 24 and sustained through week 52 (without use of rescue therapy).
Treatment-emergent adverse events (TEAEs), serious adverse events (SAEs), adverse events of special interest (AESIs), abnormalities in laboratory values, anti-drug antibody | over the entire study period (up to Week 58)
  AEs that develop or worsen or became serious during the treatment period (from first dose to 60 days after last dose).
Corticosteroid-free remission at Week 52 | at Week 52
  Remission, without receipt of systemic corticosteroids (CS) or rescue treatment within 7 days prior to the assessment time point.
Remission at Week 24 | at Week 24
  Achievement of remission at Week 24.
Time in remission through Week 52 | through Week 52
  The duration (in days) in remission to first PMR flare, up to Week 52.
Incidence rate of flare through Week 52 | through Week 52
  The number of flares and raw incidence rate over the 52-week treatment period.
Change from baseline in PMR activity score and its components at Weeks 24 and 52 | at Weeks 24 and 52
  PMR activity score is a composite score based on serum inflammatory markers, physician's global assessment of disease activity visual analog scale (VAS), patient's assessment of pain visual analog score (VAS), morning stiffness and shoulder range of motion.
Changes from baseline at Weeks 24 and 52 in the physical component summary and mental component summary from Short-form 36-item questionnaire (SF-36v2) | at Weeks 24 and 52
  The SF-36v2 yields scores for eight domains (Physical Functioning, Role-Physical, Bodily pain, General health, Vitality, Social Functioning, Role-Emotional, and Mental Health), as well as 2 standardized summary scores - the physical component summary (PCS) and mental component summary (MCS).

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org